CLINICAL TRIAL: NCT01732289
Title: Genetic Study of Age Related Hearing Loss
Acronym: ARHL
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Clinical professor, National Taiwan University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 200806069R; Taiwan NSC 97-2314-B-002-107
Record Dates: First submitted 2008-09-01; First posted 2012-11-22 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Age-related Hearing Loss; Presbycusis
Keywords: Age-related hearing loss; Gene; Single nucleotide polymorphism; environmental factors
MeSH Terms: conditions — Presbycusis | interventions — Genes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Genetic: genes

INTERVENTIONS:
Genetic: genes — Draw blood for genetic screening
  Other Names: no other name

SUMMARY:
Age-related hearing loss, or presbyacusis, is one of the most common chronically handicapped conditions for the elderly. Many factors including genetics, diet, diseases, drugs, socioeconomic factors and environmental variables were considered to be related to the development of presbyacusis. Evidences have shown that genetic factors play an important role on presbyacusis. However, which genes or their genotypes are associated with presbycusis remain unknown.

The aim of this project was to evaluate the association between the genotype of candidate genes and presbyacusis by cross-section and case-control study. In the first stage, the investigators plan to select 700 healthy subjects older than 50 with symmetric, sensorineural hearing loss. The subjects will receive basic otologic examination, pure tone audiometry, questionnaire, and genotype analysis. Because gender and age would affect hearing loss significantly, The investigators will convert the hearing level of all subjects into a gender and age independent Z-score according to ISO 7029 standard. And, The investigators define subjects within higher 30 % of Z-score as the presbyacusis group, and subjects within lower 30% of Z-score as the control group. Finally, The investigators perform Chi square analysis to test the association between genotype of candidate genes or their combinations in both groups, and calculate the odds ratio for presbyacusis between different genotype of candidate genes. Further more, we will evaluate the effect of genotype of candidate genes, environment factors, and gene-environmental interaction on the severity of presbyacusis by multivariate logistic regression.

In the second stage, The investigators wish to know the pattern of genotype and hearing level in the high risk families, according to results from the first stage, by description and case-control study. The investigators will perform t-test to evaluate the difference of Z-score in both groups. Besides, The investigators try to evaluate the effects of genotypes, environment factors, and gene-environmental interaction on hearing level in high risk families by multivariate logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged 45 or above, both male and female came to the hospital for health check up

Exclusion Criteria:

* known ontological disease age under 45 noise exposure history history of ototoxicity psychiatric diseases

Min Age: 45 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2008-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
which gene or Single nucleotide polymorphism is related to age related hearing loss | 2008-2009

SECONDARY OUTCOMES:
Which environmental factor(s) or systemic diseases are related to age related hearing loss | 2008-2009

CONTACTS AND LOCATIONS:
Overall Officials: Tien-Chen Liu, MD, PhD, Principal Investigator — Department of Otolayrngology, National Taiwan Univserity Hospital
Locations (1):
- National Taiwna University Hospital, Taipei, Taiwan